CLINICAL TRIAL: NCT06824714
Title: A Prospective, Observational Study on Prediction of Risk of Vascular Structural Damage in Patients With Large Vessel Vasculitis(LVV) Based on PET/MRA Image Evaluation System
Brief Title: Prediction of Risk of Vascular Structural Damage in Patients With Large Vessel Vasculitis (LVV) Based on PET/MRA Image Evaluation System
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Rui LIU, MD, MD, Nanjing Medical University
Other Study IDs: 2024-SR-693
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Large Vessel Vasculitis
Keywords: Large Vessel Vasculitis; PET; MRA; SUVmax; TBA
MeSH Terms: interventions — Glucocorticoids; Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clinically suspected or confirmed large vessel vasculitis (LVV)
  Interventions: Drug: glucocorticoid, immunosuppressants, targeted therapy

INTERVENTIONS:
Drug: glucocorticoid, immunosuppressants, targeted therapy — Drug intervention protocol will be determined by clinicians

SUMMARY:
Large vessel vasculitis (LVV) causes vascular inflammation, leading to serious complications such as aneurysm formation and stroke. It is difficult to identify the inflammation of the vessel wall by the current imaging methods, thus affecting the timing of treatment and selection of treatment options. Improved examination methods to determine disease activity are highly needed to guide treatment.

DETAILED DESCRIPTION:
This study was designed to assess vascular wall inflammation in patients with large vessel vasculitis by positron emission tomography and magnetic resonance imaging (PET/MRA). The study has a 12-month follow-up period. After completing the baseline clinical assessment, laboratory test and PET/MRA assessment, the intervention protocol will be determined by clinicians. The patients will visit the clinic every 1-2 months according to their specific conditions. Clinical assessment, laboratory test and PET/MRA re-examination will be completed at 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically suspected or confirmed LVV and willing to undergo PET/MRA
2. Compliance with long-term follow-up
3. Sign informed consent.

Exclusion Criteria:

1. Patients with other serious cardiovascular and cerebrovascular diseases, malignant tumors, infectious diseases, severe renal insufficiency.
2. Severe mental disorders, severe claustrophobia unable to cooperate with the examination.
3. Patients equipped with cardiac pacemaker, artificial heart valve, ferromagnetic vascular clamp after vascular surgery, aneurysm clamp, artificial cochlea, insulin pump and other drug dosage control devices, steel nail plate and other metal internal fixation, artificial joint, electronic eye, artificial eye.
4. Allergic to contrast medium.
5. Pregnant or lactating women.

Withdrawal criteria:

1. Any exclusion criteria emerged during patient follow-up.
2. Voluntarily withdrew from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically suspected or confirmed LVV
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Vascular structural progression | 12 months
  Vascular structural progression indicated by PET/MRA (including new vessel wall thickening, increased thickening, vascular stenosis or occlusion, aneurysm formation)

SECONDARY OUTCOMES:
SUV max | 12 months
  Standardized uptake values（SUV） is a semiquantitative measurement of tumor uptake of FDG derived by measuring the ratio of radioactivity in the tumor to the expected baseline activity in the body. The SUVmax is defined as the maximum value for SUV in a Volume of interest (VOI) representing the highest metabolism in the tumor.
TBA | 12 months
  A template-based approach (TBA) consists in matching a model to the patient's anatomy so that the known attenuation map from the model can be applied to the patient data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology and Immunology, Jiangsu Province Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez-Moller A, Nekolla SG. Attenuation correction for PET/MR: problems, novel approaches and practical solutions. Z Med Phys. 2012 Dec;22(4):299-310. doi: 10.1016/j.zemedi.2012.08.003. Epub 2012 Aug 25. PMID 22925653
- [Background] Kostakoglu L, Chauvie S. Metabolic Tumor Volume Metrics in Lymphoma. Semin Nucl Med. 2018 Jan;48(1):50-66. doi: 10.1053/j.semnuclmed.2017.09.005. PMID 29195618